CLINICAL TRIAL: NCT03103997
Title: Wet Heparinized Suction: A Novel Technique to Enhance Tissue Acquisition for Endoscopic Ultrasound Guided Liver Biopsy (EUS-LB): A Prospective Trial
Brief Title: Wet Heparin for Obtaining Liver Tissue for EUS Guided Liver Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2016-0300
Record Dates: First submitted 2017-03-14; First posted 2017-04-07 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Liver Diseases
Keywords: Liver; EUS; Biopsy; Heparin
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Intervention Model Description: Subjects enrolled will undergo EUS-guided biopsies in the following manner. First pass needle out of package without preparation and full suction. Second pass: needle flushed with heparin, then flushed with air and suction, dry heparin. Third pass: needle flushed with heparin and then 2 cc of liquid added to suction syringe and attached, wet heparin.
Who Masked: Outcomes Assessor
Masking Description: Participants undergo each biopsy in the protocol. The care provider will be directing and performing each needle pass. The outcome assessor will be unaware of each group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- New Needle (Active Comparator): EUS-guided liver biopsy with needle and suction, no preparation
  Interventions: Procedure: EUS-guided liver biopsy
- Dry Heparin (Experimental): EUS-guided liver biopsy with needle flushed with heparin, then flushed with air, suction then attached
  Interventions: Procedure: EUS-guided liver biopsy
- Wet Heparin (Experimental): EUS-guided liver biopsy with needle flushed with heparin, 2 cc of liquid added to suction then attached.
  Interventions: Procedure: EUS-guided liver biopsy

INTERVENTIONS:
Procedure: EUS-guided liver biopsy — EUS-guided liver biopsy using needles with various preparations

SUMMARY:
Since its inception, endoscopic ultrasound with fine needle aspiration (EUS-FNA) has proven a valuable diagnostic and prognostic tool for evaluating a diverse number of pathologies. One such pathology is chronic liver disease (CLD), for which EUS-guided liver biopsy has become a well-accepted method for tissues acquisition. EUS-LB also been compared with percutaneous and transguluar routes showing at least comparable ability to obtain adequate tissue for CLD.

Though enhancements to EUS-FNA, such as dry suction, stylet pull have not proven to demonstrate increased diagnostic accuracy for EUS-FNA, the use of wet suction technique (WEST) has demonstrated the ability to obtain more cellular tissue samples with less blood contamination. In an attempt to obtain further improvement in tissue adequacy, with less blood contamination for EUS-LB, the use of wet heparinized needles will be investigated as compared with conventional EUS-LB for patients with CLD. To do this subjects shall be selected to undergo EUS-LB. As it is the standard to perform 3 needle passes during EUS-LB, subjects will undergo one pass with the following designations: pass 1: conventional EUS-LB [no flush], pass 2: dry heparin heparin [5 milliliters (mL) of heparin flushed and then flushed with air], and pass 3: wet heparin [5 milliliters (mL) of heparin flushed and retained in the needle]. It is predicted that specimens collected with heparinized needle shall show improved adequacy compared with conventional EUS-LB. It is also predicted that the heparin wash will lead to less blood contamination compared with conventional methods. Subjects shall also be monitored for adverse events (AE).

DETAILED DESCRIPTION:
3 BACKGROUND AND SIGNIFICANCE Since its inception in 1992, endoscopic ultrasound with fine needle aspiration (EUS-FNA) has continued to be an evolving method for obtaining diagnostically accuracy for gastrointestinal, and extra-luminal pathology. Present society guidelines by both the European Society of Gastrointestinal Endoscopy (ESGE) and American Society of Gastrointestinal Endoscopy (ASGE) have estimated an overall 60-90% diagnostic accuracy of EUS-FNA. However, this accuracy is dependent upon determination of adequacy by expert gastrointestinal pathologists, which may not be available at all centers.

To enhance the diagnostic accuracy of EUS-FNA, several techniques have been described including, acquisition of a core specimen by fine needle biopsy (FNB), the use of a stylet, and suction. Regarding FNB, this technique allows for acquisition of a tissue specimen with intact tissue architecture and therefore more ability for immunohistochemical staining (IHC). The original generations of FNB needles have been studies, demonstrating no noticeable advantage of convention FNA. More recent evolutions of these FNB needles have led to promising preliminary results. For obtaining EUS-guided liver biopsy (EUS-LB), the technical success was 100% and over 91% diagnostic accuracy. Furthermore, EUS-LB appears to have a higher diagnostic accuracy for chronic liver disease (CLD) compared with percutaneous (PLB) and transgulular (TLB) routes. Overall, EUS-FNB appears to be a promising additional to EUS guided tissue acquisition, which shall lead to improved diagnostic accuracy.

In addition to EUS-FNB, both EUS-FNA with stylet use and suction, have gained some notoriety. It is important to note that there is no definitive evidence of improved diagnostic accuracy of EUS-FNA with these methods. One caveat to these supplemental methods for EUS-FNA, would be the use of "wet suction" technique (WEST) for EUS-FNA. The wet suction technique involved the use of 5 milliliters (mL) of 0.9% normal saline (NS) to supplant the traditional column of air present in the FNA needle. When compared to traditional EUS-FNA, the WEST demonstrated an increase in cellularity of the cellblock, improved specimen accuracy and no difference in the blood contamination compared with standard EUS-FNA. Though not specifically an EUS technique, using heparinized needles for PLB of liver lesions, has been described as well. Despite these promising results, this technique has never been employed as an enhancement to EUS-FNA.

Therefore in this study a heparinized solution (wet heparin) shall be employed for the acquisition of tissue in EUS-LB compared with dry heparin and convention EUS-LB. It is predicted that EUS-LB wet heparin will lead to less blood contamination and more adequate tissue acquisition, as compared with dry heparin and conventional EUS-LB.

Primary End Points

1. Proportion of cases for which a histologic diagnosis could be made based upon the amount of tissue obtained with the needle.
2. Number of portal tracts (PT) in the specimen
3. Aggregate specimen length (ASL), length of the longest piece (LLP), and degree of fragmentation Secondary End Points

1. Presence of a visible core specimen 2. Presence of visible clots in specimen 3. Adverse events (AE) and serious adverse events (SAE) 4 HYPOTHESIS AND SPECIFIC AIMS 4.1 Hypothesis It is predicted that EUS-LB with wet heparin will lead to less blood contamination and more adequate tissue acquisition, as compared with dry heparin and conventional EUS-LB 4. 2 Specific Aim 1 To determine the adequacy of EUS-LB using wet and dry heparin 4.3 Specific Aim 2 To determine the degree of blood contamination for EUS-LB using wet heparin and dry heparin 4.4 Specific Aim 3 To determine the adequacy for EUS-LB using wet heparin and dry heparin 5 PRELIMINARY DATA Heparin flush has been used previously in several patients undergoing EUS-guided liver biopsy, and cores of liver tissue can be obtained. It has been found that this needle preparation using heparin flush has led to the presence of less blood contamination of tissue and therefore improved diagnostic accuracy and ability to make the diagnosis.

6 STUDY DESIGN 6.1 Description This is an open-labeled, prospective trial comparing tissue acquisition adequacy and blood contamination for EUS-LB using wet heparin (Group A), dry heparin (Group B) and conventional EUS-LB (Group C).

Group A: Needle flushed with 5mL of heparin, left in the EUS-FNB needle Group B: Needle flushed with 5mL of heparin, then flushed with air to dry Group C: Needle not flushed with solution

Subjects shall then undergo EUS-LB (see below) with 3 trans-gastric passes total in the left lobe, as is the present standard of practice. Pass 1: Group C, Pass 2: Group B, Pass 3: Group A.

After EUS-LB, the tissue sample shall then be evaluated after each pass by the endosongrapher performing EUS-LB for tissue length. The tissue and fluid washed from the tissue specimens shall then be sent for processing, as described below, and evaluated for the primary and secondary outcomes by 2 expert pathologists, blinded to which arm each specimen had come from. Patients shall then receive a telephone call 7 days after EUS-LB to evaluate for adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing EUS-LB
2. Platelet count > 50,000
3. International normalized ratio (INR) < 1.5
4. Age > 18 years
5. Non-pregnant patients

Exclusion Criteria:

1. Age < 18 years
2. Pregnant Patients
3. Inability to obtain consent
4. Anticoagulants or anti-platelet agents use (excluding aspirin) within the last 7-10 days
5. Platelet count < 50,000
6. INR > 1.5
7. Presence of ascites
8. Known liver cirrhosis
9. Patients with a heparin or porcine allergy
10. Patients with prior heparin induced thrombocytopenia (HIT)
11. Patient's with religious aversion to porcine-containing products

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of cases for which a histologic diagnosis could be made based upon Proportion of cases for which a histologic diagnosis could be made based upon the amount of tissue obtained with the needle | 7 days
  Proportion of cases for which a histologic diagnosis could be made based upon the amount of tissue obtained with the needle

SECONDARY OUTCOMES:
The Number of patients with a visible core after needle biopsy | Presence of a visible core specimen (yes/no) at time 7 days
  Day of Procedure
The Number of patients with a visible clot after needle biopsy | Presence of visible clots in specimen (yes/no) at time 7 days
  Day of Procedure
The Number of patients with visible bleeding after needle biopsy | 7 Days
  Patient with blood visible from patient's mouth, rectum with a 2 gram drop in hemoglobin
The Number of patients with Pain 1 Day after needle biopsy | 1 Days
  Pain using Likert score 0-10 (10 worst)
The Number of patients with Pain 7 Day after needle biopsy | 7 Days
  Pain using Likert score 0-10 (10 worst)
The Number of patients requiring medical care after needle biopsy | 7 Days
  Patient requiring visit to healthcare center (emergency room, hospital, call to service) within time 7 days
Number of portal tracts (PT) in the specimen (total) under histologic examination | 7 Days
  Number of portal tracts (PT) in the specimen (total) under histologic examination
Aggregate Specimen Length under histologic examination | 7 Days
  Length of all the tissue (centimeters) by adding the sum of all pieces
Length of the longest piece under histologic examination | 7 Days
  length of the longest tissue biopsy piece (centimeters) as measured by pathology

CONTACTS AND LOCATIONS:
Overall Officials: David L Diehl, M.D., Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Medical Center, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vilmann P, Jacobsen GK, Henriksen FW, Hancke S. Endoscopic ultrasonography with guided fine needle aspiration biopsy in pancreatic disease. Gastrointest Endosc. 1992 Mar-Apr;38(2):172-3. doi: 10.1016/s0016-5107(92)70385-x. No abstract available. PMID 1568614
- [Result] Dumonceau JM, Polkowski M, Larghi A, Vilmann P, Giovannini M, Frossard JL, Heresbach D, Pujol B, Fernandez-Esparrach G, Vazquez-Sequeiros E, Gines A; European Society of Gastrointestinal Endoscopy. Indications, results, and clinical impact of endoscopic ultrasound (EUS)-guided sampling in gastroenterology: European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2011 Oct;43(10):897-912. doi: 10.1055/s-0030-1256754. Epub 2011 Aug 12. PMID 21842456
- [Result] Hebert-Magee S, Bae S, Varadarajulu S, Ramesh J, Frost AR, Eloubeidi MA, Eltoum IA. The presence of a cytopathologist increases the diagnostic accuracy of endoscopic ultrasound-guided fine needle aspiration cytology for pancreatic adenocarcinoma: a meta-analysis. Cytopathology. 2013 Jun;24(3):159-71. doi: 10.1111/cyt.12071. PMID 23711182
- [Result] Iglesias-Garcia J, Dominguez-Munoz JE, Abdulkader I, Larino-Noia J, Eugenyeva E, Lozano-Leon A, Forteza-Vila J. Influence of on-site cytopathology evaluation on the diagnostic accuracy of endoscopic ultrasound-guided fine needle aspiration (EUS-FNA) of solid pancreatic masses. Am J Gastroenterol. 2011 Sep;106(9):1705-10. doi: 10.1038/ajg.2011.119. Epub 2011 Apr 12. PMID 21483464
- [Result] Eloubeidi MA, Tamhane A, Jhala N, Chhieng D, Jhala D, Crowe DR, Eltoum IA. Agreement between rapid onsite and final cytologic interpretations of EUS-guided FNA specimens: implications for the endosonographer and patient management. Am J Gastroenterol. 2006 Dec;101(12):2841-7. doi: 10.1111/j.1572-0241.2006.00852.x. Epub 2006 Oct 6. PMID 17026562
- [Result] Jhala NC, Jhala DN, Chhieng DC, Eloubeidi MA, Eltoum IA. Endoscopic ultrasound-guided fine-needle aspiration. A cytopathologist's perspective. Am J Clin Pathol. 2003 Sep;120(3):351-67. doi: 10.1309/MFRF-J0XY-JLN8-NVDP. PMID 14502798
- [Result] Harada N, Kouzu T, Arima M, Isono K. Endoscopic ultrasound-guided histologic needle biopsy: preliminary results using a newly developed endoscopic ultrasound transducer. Gastrointest Endosc. 1996 Sep;44(3):327-30. doi: 10.1016/s0016-5107(96)70173-6. No abstract available. PMID 8885355
- [Result] Binmoeller KF, Thul R, Rathod V, Henke P, Brand B, Jabusch HC, Soehendra N. Endoscopic ultrasound-guided, 18-gauge, fine needle aspiration biopsy of the pancreas using a 2.8 mm channel convex array echoendoscope. Gastrointest Endosc. 1998 Feb;47(2):121-7. doi: 10.1016/s0016-5107(98)70343-8. PMID 9512275
- [Result] Voss M, Hammel P, Molas G, Palazzo L, Dancour A, O'Toole D, Terris B, Degott C, Bernades P, Ruszniewski P. Value of endoscopic ultrasound guided fine needle aspiration biopsy in the diagnosis of solid pancreatic masses. Gut. 2000 Feb;46(2):244-9. doi: 10.1136/gut.46.2.244. PMID 10644320
- [Result] Varadarajulu S, Fraig M, Schmulewitz N, Roberts S, Wildi S, Hawes RH, Hoffman BJ, Wallace MB. Comparison of EUS-guided 19-gauge Trucut needle biopsy with EUS-guided fine-needle aspiration. Endoscopy. 2004 May;36(5):397-401. doi: 10.1055/s-2004-814316. PMID 15100946
- [Result] Shah SM, Ribeiro A, Levi J, Jorda M, Rocha-Lima C, Sleeman D, Hamilton-Nelson K, Ganjei-Azar P, Barkin J. EUS-guided fine needle aspiration with and without trucut biopsy of pancreatic masses. JOP. 2008 Jul 10;9(4):422-30. PMID 18648133
- [Result] Thomas T, Kaye PV, Ragunath K, Aithal G. Efficacy, safety, and predictive factors for a positive yield of EUS-guided Trucut biopsy: a large tertiary referral center experience. Am J Gastroenterol. 2009 Mar;104(3):584-91. doi: 10.1038/ajg.2008.97. Epub 2009 Feb 10. PMID 19262518
- [Result] Levy MJ, Jondal ML, Clain J, Wiersema MJ. Preliminary experience with an EUS-guided trucut biopsy needle compared with EUS-guided FNA. Gastrointest Endosc. 2003 Jan;57(1):101-6. doi: 10.1067/mge.2003.49. PMID 12518144
- [Result] Iglesias-Garcia J, Poley JW, Larghi A, Giovannini M, Petrone MC, Abdulkader I, Monges G, Costamagna G, Arcidiacono P, Biermann K, Rindi G, Bories E, Dogloni C, Bruno M, Dominguez-Munoz JE. Feasibility and yield of a new EUS histology needle: results from a multicenter, pooled, cohort study. Gastrointest Endosc. 2011 Jun;73(6):1189-96. doi: 10.1016/j.gie.2011.01.053. Epub 2011 Mar 21. PMID 21420083
- [Result] Larghi A, Iglesias-Garcia J, Poley JW, Monges G, Petrone MC, Rindi G, Abdulkader I, Arcidiacono PG, Costamagna G, Biermann K, Bories E, Doglioni C, Dominguez-Munoz JE, Hassan C, Bruno M, Giovannini M. Feasibility and yield of a novel 22-gauge histology EUS needle in patients with pancreatic masses: a multicenter prospective cohort study. Surg Endosc. 2013 Oct;27(10):3733-8. doi: 10.1007/s00464-013-2957-9. Epub 2013 May 4. PMID 23644834
- [Result] Bang JY, Hebert-Magee S, Trevino J, Ramesh J, Varadarajulu S. Randomized trial comparing the 22-gauge aspiration and 22-gauge biopsy needles for EUS-guided sampling of solid pancreatic mass lesions. Gastrointest Endosc. 2012 Aug;76(2):321-7. doi: 10.1016/j.gie.2012.03.1392. Epub 2012 May 31. PMID 22658389
- [Result] Iwashita T, Nakai Y, Samarasena JB, Park DH, Zhang Z, Gu M, Lee JG, Chang KJ. High single-pass diagnostic yield of a new 25-gauge core biopsy needle for EUS-guided FNA biopsy in solid pancreatic lesions. Gastrointest Endosc. 2013 Jun;77(6):909-15. doi: 10.1016/j.gie.2013.01.001. Epub 2013 Feb 20. PMID 23433596
- [Result] Stavropoulos SN, Im GY, Jlayer Z, Harris MD, Pitea TC, Turi GK, Malet PF, Friedel DM, Grendell JH. High yield of same-session EUS-guided liver biopsy by 19-gauge FNA needle in patients undergoing EUS to exclude biliary obstruction. Gastrointest Endosc. 2012 Feb;75(2):310-8. doi: 10.1016/j.gie.2011.09.043. PMID 22248599
- [Result] Gor N, Salem SB, Jakate S, Patel R, Shah N, Patil A. Histological adequacy of EUS-guided liver biopsy when using a 19-gauge non-Tru-Cut FNA needle. Gastrointest Endosc. 2014 Jan;79(1):170-2. doi: 10.1016/j.gie.2013.06.031. Epub 2013 Jul 31. No abstract available. PMID 23916397
- [Result] Diehl DL, Johal AS, Khara HS, Stavropoulos SN, Al-Haddad M, Ramesh J, Varadarajulu S, Aslanian H, Gordon SR, Shieh FK, Pineda-Bonilla JJ, Dunkelberger T, Gondim DD, Chen EZ. Endoscopic ultrasound-guided liver biopsy: a multicenter experience. Endosc Int Open. 2015 Jun;3(3):E210-5. doi: 10.1055/s-0034-1391412. Epub 2015 Feb 27. PMID 26171433
- [Result] DeWitt J, LeBlanc J, McHenry L, Ciaccia D, Imperiale T, Chappo J, Cramer H, McGreevy K, Chriswell M, Sherman S. Endoscopic ultrasound-guided fine needle aspiration cytology of solid liver lesions: a large single-center experience. Am J Gastroenterol. 2003 Sep;98(9):1976-81. doi: 10.1111/j.1572-0241.2003.07638.x. PMID 14499774
- [Result] Hollerbach S, Willert J, Topalidis T, Reiser M, Schmiegel W. Endoscopic ultrasound-guided fine-needle aspiration biopsy of liver lesions: histological and cytological assessment. Endoscopy. 2003 Sep;35(9):743-9. doi: 10.1055/s-2003-41593. PMID 12929021
- [Result] tenBerge J, Hoffman BJ, Hawes RH, Van Enckevort C, Giovannini M, Erickson RA, Catalano MF, Fogel R, Mallery S, Faigel DO, Ferrari AP, Waxman I, Palazzo L, Ben-Menachem T, Jowell PS, McGrath KM, Kowalski TE, Nguyen CC, Wassef WY, Yamao K, Chak A, Greenwald BD, Woodward TA, Vilmann P, Sabbagh L, Wallace MB. EUS-guided fine needle aspiration of the liver: indications, yield, and safety based on an international survey of 167 cases. Gastrointest Endosc. 2002 Jun;55(7):859-62. doi: 10.1067/mge.2002.124557. PMID 12024141
- [Result] Pineda JJ, Diehl DL, Miao CL, Johal AS, Khara HS, Bhanushali A, Chen EZ. EUS-guided liver biopsy provides diagnostic samples comparable with those via the percutaneous or transjugular route. Gastrointest Endosc. 2016 Feb;83(2):360-5. doi: 10.1016/j.gie.2015.08.025. Epub 2015 Aug 22. PMID 26301407
- [Result] Wallace MB, Kennedy T, Durkalski V, Eloubeidi MA, Etamad R, Matsuda K, Lewin D, Van Velse A, Hennesey W, Hawes RH, Hoffman BJ. Randomized controlled trial of EUS-guided fine needle aspiration techniques for the detection of malignant lymphadenopathy. Gastrointest Endosc. 2001 Oct;54(4):441-7. doi: 10.1067/mge.2001.117764. PMID 11577304
- [Result] Sahai AV, Paquin SC, Gariepy G. A prospective comparison of endoscopic ultrasound-guided fine needle aspiration results obtained in the same lesion, with and without the needle stylet. Endoscopy. 2010 Nov;42(11):900-3. doi: 10.1055/s-0030-1255676. Epub 2010 Aug 19. PMID 20725886
- [Result] Rastogi A, Wani S, Gupta N, Singh V, Gaddam S, Reddymasu S, Ulusarac O, Fan F, Romanas M, Dennis KL, Sharma P, Bansal A, Oropeza-Vail M, Olyaee M. A prospective, single-blind, randomized, controlled trial of EUS-guided FNA with and without a stylet. Gastrointest Endosc. 2011 Jul;74(1):58-64. doi: 10.1016/j.gie.2011.02.015. Epub 2011 Apr 23. PMID 21514932
- [Result] Wani S, Gupta N, Gaddam S, Singh V, Ulusarac O, Romanas M, Bansal A, Sharma P, Olyaee MS, Rastogi A. A comparative study of endoscopic ultrasound guided fine needle aspiration with and without a stylet. Dig Dis Sci. 2011 Aug;56(8):2409-14. doi: 10.1007/s10620-011-1608-z. Epub 2011 Feb 17. PMID 21327919
- [Result] Puri R, Vilmann P, Saftoiu A, Skov BG, Linnemann D, Hassan H, Garcia ES, Gorunescu F. Randomized controlled trial of endoscopic ultrasound-guided fine-needle sampling with or without suction for better cytological diagnosis. Scand J Gastroenterol. 2009;44(4):499-504. doi: 10.1080/00365520802647392. PMID 19117242
- [Result] Attam R, Arain MA, Bloechl SJ, Trikudanathan G, Munigala S, Bakman Y, Singh M, Wallace T, Henderson JB, Catalano MF, Guda NM. "Wet suction technique (WEST)": a novel way to enhance the quality of EUS-FNA aspirate. Results of a prospective, single-blind, randomized, controlled trial using a 22-gauge needle for EUS-FNA of solid lesions. Gastrointest Endosc. 2015;81(6):1401-7. doi: 10.1016/j.gie.2014.11.023. Epub 2015 Feb 27. PMID 25733127
- [Result] Kasugai H, Yamamoto R, Tatsuta M, Okano Y, Okuda S, Kishigami Y, Kitamura T, Wada A, Tamura H. Value of heparinized fine-needle aspiration biopsy in liver malignancy. AJR Am J Roentgenol. 1985 Feb;144(2):243-4. doi: 10.2214/ajr.144.2.243. PMID 2981458
- [Result] Colloredo G, Guido M, Sonzogni A, Leandro G. Impact of liver biopsy size on histological evaluation of chronic viral hepatitis: the smaller the sample, the milder the disease. J Hepatol. 2003 Aug;39(2):239-44. doi: 10.1016/s0168-8278(03)00191-0. PMID 12873821
- [Result] Crawford AR, Lin XZ, Crawford JM. The normal adult human liver biopsy: a quantitative reference standard. Hepatology. 1998 Aug;28(2):323-31. doi: 10.1002/hep.510280206. PMID 9695993
- [Result] Rocken C, Meier H, Klauck S, Wolff S, Malfertheiner P, Roessner A. Large-needle biopsy versus thin-needle biopsy in diagnostic pathology of liver diseases. Liver. 2001 Dec;21(6):391-7. doi: 10.1034/j.1600-0676.2001.210605.x. PMID 11903883
- [Result] Bhatia V, Hijioka S, Hara K, Mizuno N, Imaoka H, Yamao K. Endoscopic ultrasound description of liver segmentation and anatomy. Dig Endosc. 2014 May;26(3):482-90. doi: 10.1111/den.12216. Epub 2013 Dec 19. PMID 24355092
- [Result] ASGE Standards of Practice Committee; Early DS, Acosta RD, Chandrasekhara V, Chathadi KV, Decker GA, Evans JA, Fanelli RD, Fisher DA, Fonkalsrud L, Hwang JH, Jue TL, Khashab MA, Lightdale JR, Muthusamy VR, Pasha SF, Saltzman JR, Sharaf RN, Shergill AK, Cash BD. Adverse events associated with EUS and EUS with FNA. Gastrointest Endosc. 2013 Jun;77(6):839-43. doi: 10.1016/j.gie.2013.02.018. No abstract available. PMID 23684089
- [Result] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503
- [Derived] Mok SRS, Diehl DL, Johal AS, Khara HS, Confer BD, Mudireddy PR, Kirchner HL, Chen ZE. A prospective pilot comparison of wet and dry heparinized suction for EUS-guided liver biopsy (with videos). Gastrointest Endosc. 2018 Dec;88(6):919-925. doi: 10.1016/j.gie.2018.07.036. Epub 2018 Aug 16. PMID 30120956